CLINICAL TRIAL: NCT01667653
Title: A Randomized Parallel Group Study to Evaluate the Effect of a Probiotic Product in Healthy Adults Undergoing Antibiotic Treatment
Brief Title: Probiotic Product in Healthy Adults Undergoing Antibiotic Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Danisco (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11PDHD
Record Dates: First submitted 2012-03-23; First posted 2012-08-17 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Antibiotic Therapy
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Augmentin/Probiotic (Experimental): Participants are provided in double blinded fashion probiotic to take with antibiotics
  Interventions: Dietary Supplement: Probiotic
- Augmentin/placebo (Experimental): Participants are provided in double blinded fashion placebo to take with antibiotics
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic capsule once daily
  Arms: Augmentin/Probiotic
Dietary Supplement: Placebo — Placebo capsule once daily
  Arms: Augmentin/placebo

SUMMARY:
This is randomized, double-blind, placebo controlled, single centre; 21 days phase II clinical trial on healthy volunteers. Following baseline visit at the day of randomization, treatment with Augmentin 875mg for 7 days will be given. Concurrently and after antibiotic treatment subjects will also receive the study treatment, either probiotic or placebo. Daily Bowel Habit Diary will be completed by the subjects. The subjects will be asked to collect fecal samples for microbiological examination. The primary objective of the study is to evaluate the maintenance of intestinal microbiota composition during antibiotic treatment with Augmentin 875mg. Secondary objectives will be to evaluate the reduction in side effects associated with antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 50 years.
* Healthy as determined by laboratory results, medical history and physical exam
* Willing to give voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Body mass index ≥ 30 kg/m2
* Average number of formed bowel movements > 3 per day or < 3 per week
* Smokers
* Participation in a clinical research trial within 30 days prior to randomization
* Use of antibiotics within 60 days prior to randomization.
* Habitual use of pro- and/or prebiotic products.
* Follows a vegetarian or vegan diet
* Unstable medical conditions
* Any evidence of acute or chronic gastrointestinal disorder
* Alcohol use > 2 standard alcoholic drinks per day and/or alcohol or drug abuse within past year
* Allergy or sensitivity to test product ingredients or antibiotic
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maintenance of intestinal microbiotic composition before, during and after antibiotic treatment with Augmentin 875mg | 3 weeks
  Fecal samples collected during the 3 week period and stored frozen until analyses. Bacterial DNA is extracted from the samples and the microbial composition is analysed by molecular methods such as quantitative PCR.

SECONDARY OUTCOMES:
The influence of probiotics on side effects associated with antibiotic use | 3-weeks
  Questionaire is used to assess the tolerability of the probiotic supplementation, Bowel habit scores, adverse effects,

CONTACTS AND LOCATIONS:
Locations (1):
- KGK Synergize Inc., London/Ontario, Canada